CLINICAL TRIAL: NCT06882772
Title: Butyric Acid Supplementation for Gut Improvement After Cardiac Surgery in Kids, A Phase IIa Clinical Trial
Brief Title: Butyric Acid Supplementation for Gut Improvement After Cardiac Surgery in Kids
Acronym: BASICS-Kids
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 0839-24-FB; 11543 (Other Grant/Funding Number: Gerber Foundation)
Record Dates: First submitted 2025-02-05; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Congenital Heart Disease (CHD)
Keywords: Congenital Heart Disease; Gut Health; Microbiome; Gut Barrier Function; Inflammation
MeSH Terms: conditions — Heart Defects, Congenital; Inflammation | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 2 mL SunButyrate-TG (Arm1) (Experimental): Participants will receive 2 milliliter (mL) SunButyrate-TG once daily for 3 weeks prior to cardiac surgery.
  Interventions: Drug: 2 mL SunButyrate-TG
- 4 mL SunButyrate-TG (Arm 2) (Experimental): Participants will receive 4 milliliter (mL) SunButyrate-TG once daily for 3 weeks prior to cardiac surgery.
  Interventions: Drug: 4 mL SunButyrate-TG
- Placebo Comparator (Arm 3) (Placebo Comparator): Participants will receive either 2 milliliter (mL) or 4 mL of an inactive oil-based placebo once daily for 3 weeks prior to cardiac surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 2 mL SunButyrate-TG — Participants randomized into the 2 milliliter (mL) SunButyrate-TG will take the supplement once daily for 3 weeks prior to cardiac surgery.
  Note: This is a Dietary Supplement, but the FDA requires an Investigational New Drug (IND) number because inflammation is being treated.
  Other Names: Butyrate Liquid Supplement
  Arms: 2 mL SunButyrate-TG (Arm1)
Drug: Placebo — Participants randomized into the Placebo arm will take the oil-based placebo once daily for 3 weeks prior to cardiac surgery
  Other Names: sugar pill
  Arms: Placebo Comparator (Arm 3)
Drug: 4 mL SunButyrate-TG — Participants randomized into the 4 mL SunButyrate-TG arm will take the supplement once daily for 3 weeks prior to cardiac surgery.
  Note: This is a Dietary Supplement, but the FDA requires an Investigational New Drug (IND) number because inflammation is being treated.
  Other Names: Butyrate Liquid Supplement
  Arms: 4 mL SunButyrate-TG (Arm 2)

SUMMARY:
Butyric acid has been shown to promote gut health and improve the microbiome in multiple adult studies. In preliminary studies in older children with inflammatory bowel disease, butyric acid was shown to be safe. However, it's suitability for infants and young children with congenital heart disease (CHD) has yet to be determined.

This study will examine butyric acid supplementation in infants and children, ages 1 month to 3 years, with CHD who require cardiac surgery with cardiopulmonary bypass. Study goals include determining the safety and tolerability of butyric acid supplementation before cardiac surgery, and to identify changes in gut microbial communities, metabolic profile, and genetic markers intestinal function. Also, the study seeks to establish a reduction in inflammation (inflammatory signaling) after cardiopulmonary bypass (CPB) in participants receiving butyric acid.

DETAILED DESCRIPTION:
The goal of this study is to supplement a liquid form of butyric acid once daily for 3 weeks prior to cardiac surgery for infants and children, ages 1 month to 3 years, with congenital heart disease to improve their pre-operative gut microbiome in efforts to reduce post-operative gut permeability and reduce post-operative inflammatory signaling.

Up to 35 participants will be enrolled in each of three arms:

* 2 mL butyric acid
* 4 mL butyric acid
* Placebo.

Participants will be asked to:

* Provide blood and stool samples (baseline, post-supplement-pre-operative, 1-hr post-op, & post-op days 1-3)
* Take either 2 mL, 4 mL or placebo once daily for 3 weeks prior to cardiac surgery
* Complete a daily log to track timing of supplement administration and any side effects or adverse events experienced

Study aims:

* Aim 1 Safety and tolerability will be measured following baseline complete blood counts, complete metabolic panel to evaluate electrolytes and organ function, along with a daily log of supplementation timing and any experienced adverse events.
* Aim 2 Modulation of gut health will be measured with stool and blood samples. Changes will be measured in the gut microbiome and metabolite profiles before and after supplementation, as well as post-operatively. Gut health will be determined by measuring plasma markers of gut barrier function before and after supplementation, as well as post-operatively.
* Aim 3 Reduction of post-operative inflammatory signaling will be measured with blood samples. Plasma cytokine levels, immune cell profiles, and inflammatory gene activation with an RNA hybridization panel will be measured pre-operatively and post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Infants and Children undergoing cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Antibiotics, surgery, or chemotherapy within the past 8 weeks
* Continuous enteral feeds before surgery
* GI pathology or intestinal surgery (excluding G-tube)
* Liver disease with elevated transaminitis or dialysis-dependent renal disease

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Combined Incidence of Adverse Events and Serious Adverse Events with Butyric Acid (SunButyrate-TG) Supplementation | 3 years
  Safety will be measured by the combined incidence of adverse events (AE) and serious adverse events (SAE). These include allergic reaction, vomiting, diarrhea, abdominal distention, infection, hospitalization, or any other concern the families report. A Data Safety Monitoring Board (DSMB) will review and catalog the incidence and severity to determine study continuation. Investigators will evaluate each AE/SAE to determine the safety of the supplement in this age and participant population. AE and SAE definitions used according to FDA regulations.
  A scoring system of 1-5 will be used to determine the severity of the AE after review by the DSMB. A cumulative score of 3 or greater will require cessation of the study for that individual. If an accumulation of 20 participants or more have a score >3 the study will be stopped. If an accumulation of SAE (score of 5) in 8 or more participants, the study will be stopped.
Tolerance of SunButyrate-TG | Baseline to 3 weeks
  Tolerance will be measured by the incidence of nausea, inability to consume the supplement, or parental concern of intolerance. The tolerance scoring metric will be used to aggregate the listed criteria into a score for each participant. Each characteristic will receive a point. If a participant has a score of 2 or greater, it will be defined as intolerance. Participant study continuation will be discussed with the family in weekly calls during the supplementation period.
Changes to White Blood Cell Count with SunButyrate-TG Supplementation | Baseline to 3 weeks
  Safety will be evaluated through measurement of the white blood cell (WBC) count of the complete blood cell (CBC) count. Investigators will evaluate changes between the pre- and post-supplementation period CBC looking at changes in WBC count to quantify the incidence of leukocytosis (WBC > 15.0 x 10^9/L) and leukopenia (WBC < 6.0 x 10^9/L) after completing the supplement and prior to the surgery. Any participant that has a WBC count higher or lower than the values stated above will be documented.
Changes to Hematocrit with SunButyrate-TG | Baseline to 3 weeks
  Investigators will measure hematocrit between pre- and post-supplement time points to determine the effect of SunButyrate-TG. Investigators will evaluate changes between the pre- and post-supplementation period complete blood count (CBC) looking at changes in of anemia (hematocrit < 29%) or polycythemia (hematocrit > 45%) after completing the supplement and prior to the surgery. Any participant that has a hematocrit higher or lower than the values stated above will be documented.
Changes in Platelets with SunButyrate-TG | Baseline to 3 weeks
  Safety will be evaluated through measurement of the white blood cell (WBC) count of the complete blood cell (CBC) count. Investigators will evaluate changes between the pre- and post-supplementation period complete blood count looking at changes in platelet (PLT) count to quantify the incidence of thrombocytopenia (PLT < 30 x 10^9/L) or thrombocythemia (PLT > 750 x 10^9/L). Any participant that has a PLT count higher or lower than the values stated above will be documented.
Changes to Renal Function (BUN, Creatinine or urine output) with SunButyrate-TG | Baseline to 4 months
  Investigators will collect blood for a comprehensive metabolic panel before and after supplementation with SunButyrate-TG. Investigators will evaluate the changes in blood urea nitrogen (BUN) and Creatinine to determine evidence of renal impairment or acute kidney injury based upon Kidney Disease: Improving Global Outcomes (KDIGO) criteria (creatinine increase 1.5-1.9 times baseline or >0.3 mg/dL increase), or urine output < 0.5 mL/kg/h for 6-12 hours (excluding overnight for potty-trained children).
Changes in Liver Function with SunButyrate-TG | Baseline to 4 months
  Investigators will collect blood and measure a comprehensive metabolic panel before and after supplementation for evidence of liver injury. Investigators will determine:
  1. Presence of acidosis (pH< 7.3)
  2. Elevation of transaminitis (AST/ALT > 3 x baseline)
  3. Elevation in INR (>2 if not on coumadin)
  4. Elevation in Bilirubin (>2 mg/dL)
  5. Elevation in alkaline phosphatase (> 2 x baseline)
  If a participant meets any one of the above criteria, this will be considered evidence of liver injury and reported.
Improvement in Gut Microbiome as Measured by Alpha Diversity, Shannon Diversity Index and Simpson Diversity Index with SunButyrate-TG Supplementation | Baseline to 4 months
  Changes to the gut microbiome will be measured before and after supplementation, as well as post-operatively. Investigators will measure improvement in alpha diversity and the number of short-chain fatty acids (SCFA) producing bacterial populations.
  An improvement will be classified by an increase in alpha diversity of measurable OTU's by 12, Shannon diversity index (increase of 0.5), and Simpson diversity index (increase of 0.08), and specific number of SCFA producing organisms by 5 OTU's compared to the placebo group.
Changes in Short-Chain Fatty Acids with SunButyrate-TG | Baseline to 4 months
  Investigators will measure metabolite profiles to evaluate the amount of short-chain fatty acids (SCFA) in the gut and plasma before and after supplementation with SunButyrate-TG. This will be classified by a statistically significant increase (p<0.05) in a list of 8 different SCFA. A positive increase in SCFA production will be classified by at least 1 SCFA being significantly increased following supplementation with SunButyrate-TG compared to the placebo group.
Gut Barrier Function after SunButyrate-TG | Baseline to 4 months
  Investigators will measure 3 plasma markers of intestinal barrier function between pre- and post-supplement, as well as post-operatively. These markers are claudin-2, claudin-3, and intestinal fatty acid binding protein (FABP2). An improvement in gut barrier will be considered if there is a statistically significant reduction in the plasma marker of any of these at the post-supplementation, or post-operative time points compared to the placebo group.

SECONDARY OUTCOMES:
Reduction of Post-Operative Cytokine Values | Pre-surgery to 4 days post-operatively
  Investigators will measure cytokine levels pre- and post-surgery to determine changes in cytokine profiles of a panel of 8 different cytokines, including TNF-alpha, IL-1, IL-4, IL-6, IL-7, IL-8, IL-10, TGF-beta and IFN-gamma). An improvement in the cytokine profile will be considered if there is a statistically significant reduction in pro-inflammatory cytokines (IL-1, TNFa, IL-6, IL-4, or IL-8, IFN-gamma) or a significant increase in anti-inflammatory cytokines (IL-10 and TGF-beta) compared to the placebo group. These cytokines are measured together and will be considered a positive improvement in cytokine profiles if at least 2 pro-inflammatory cytokine values are reduced in conjunction with an increase in IL-10 and/or TGF-beta.
Changes in Neutrophils After Surgery with SunButyrate-TG | Pre-surgery to 4 days post-operatively
  Investigators will evaluate immune cell profiles in participants before and after surgery. Investigators will evaluate shifts in neutrophils. A significant change will be considered if there is a reduction of greater than 5% total neutrophil count via flow cytometry.
Changes in Macrophages After Surgery with SunButyrate-TG | Pre-surgery to 4 days post-operatively
  Investigators will evaluate immune cell profiles in participants before and after surgery. Investigators will evaluate shifts in macrophages. A significant change will be considered if there is a reduction of greater than 5% total macrophage count via flow cytometry.
Changes in T-regulatory Cells After Surgery with SunButyrate-TG | Pre-surgery to 4 days post-operatively
  Investigators will evaluate immune cell profiles in participants before and after surgery. Investigators will evaluate shifts in T-regulatory cells (T-cell). A significant change will be considered if there is an increase of greater than 10% in T-regulatory cell count via flow cytometry.
Changes in Natural Killer T-cells Cells After Surgery with SunButyrate-TG | Pre-surgery to 4 days post-operatively
  Investigators will evaluate immune cell profiles in participants before and after surgery. Investigators will evaluate shifts in natural killer T-cells (NK T-cell). A significant change will be considered if there is a reduction of greater than 10% total NK T-cell count via flow cytometry.

OTHER OUTCOMES:
Changes in Inflammatory Gene Activation | Pre-surgery to 4 days post-operatively
  Investigators will measure inflammatory genes using an ribonucleic acid (RNA) hybridization panel and evaluate the level of activation of these genes pre-and post-surgery to determine a decrease in inflammatory signaling following supplementation with SunButyrate-TG compared to placebo. These inflammatory gene profiles are identified as a panel are are unable to be separated out. The entirety of the inflammatory gene profile will be evaluated together to assess changes in inflammatory gene activation.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Salomon, MD, MBA, Principal Investigator — University of Nebraska
Locations (1):
- Children's Nebraska, 8200 Dodge St, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant information will be partially de-identified. Information related to age, gender, ethnicity, and cardiac lesion will be shared. Additional information regarding the cardiac surgery, Society of Thoracic Surgeons-European Association for Cardio-Thoracic Surgery (STAT) category, and lab values will also be included.
Supporting Information: Study Protocol, CSR
Time Frame: Information will be shared after completion of the study starting in 2029 and be available for 5 years.
Access Criteria: Information will be shared upon request to the PI.